CLINICAL TRIAL: NCT00006247
Title: A Phase I Study of SU5416 in Pediatric Patients With Recurrent or Progressive Poor Prognosis Brain Tumors
Brief Title: SU5416 in Treating Children With Recurrent or Progressive Brain Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The pharmaceutical company discontinued further development of SU5416.
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett/PBTC Operations and Biostatistics Center Executive Director, Pediatric Brain Tumor Consortium
Purpose: Treatment
Other Study IDs: CDR0000068179; PBTC-002
Record Dates: First submitted 2000-09-11; First posted 2003-12-24 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood craniopharyngioma; childhood central nervous system germ cell tumor; childhood oligodendroglioma; childhood choroid plexus tumor; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Choroid Plexus Neoplasms; Astrocytoma; Medulloblastoma; Optic Nerve Glioma; Familial ependymoma | interventions — Semaxinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: semaxanib
  Other Names: SU5416

SUMMARY:
RATIONALE: SU5416 may stop the growth of brain cancer cells by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the safety of delivering SU5416 in children who have recurrent or progressive brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the qualitative and quantitative toxicity of SU5416 in pediatric patients with recurrent or progressive brain tumors. II. Determine the acute and chronic dose-limiting toxicity and cumulative toxicity of this regimen in these patients. III. Determine the maximum tolerated dose and pharmacokinetics of this regimen in this patient population. IV. Determine the effects of hepatic enzyme-inducing drugs, such as anticonvulsant agents, on the pharmacokinetics of this regimen in these patients. V. Determine the efficacy, in a preliminary manner, of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to concurrent use of enzyme-inducing anticonvulsant drugs (yes vs no drugs or modest-induction drugs). Patients receive SU5416 IV over 1 hour twice a week for 6 weeks. Treatment repeats every 6 weeks for 17 courses (approximately 2 years) in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients in each stratum receive escalating doses of SU5416 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 50 patients (25 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven malignant recurrent or progressive brain tumor at initial presentation or at time of recurrence or progression for which no standard curative therapy exists Histologic verification for brainstem gliomas may be waived Bone marrow involvement allowed

PATIENT CHARACTERISTICS: Age: 21 and under Performance status: Karnofsky 60-100% Life expectancy: More than 8 weeks Hematopoietic: Absolute neutrophil count greater than 1,000/mm3* Platelet count greater than 75,000/mm3* Hemoglobin greater than 9 g/dL *Transfusion independent Hepatic: Bilirubin normal for age SGOT and SGPT less than 2.5 times normal for age PT/PTT no greater than 1.2 times upper limit of normal Albumin greater than 3 g/dL No overt hepatic disease Renal: Creatinine no greater than 1.5 times normal for age OR Glomerular filtration rate greater than 70 mL/min No overt renal disease Cardiovascular: No deep venous or arterial thrombosis within the past 3 months No history of myocardial infarction, severe or unstable angina, or severe peripheral vascular disease No overt cardiac disease No prior cerebral bleeds Pulmonary: No pulmonary embolism within the past 3 months No overt pulmonary disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No known allergies to paclitaxel or other agent that uses Cremophor EL No uncontrolled infection Neurological deficits allowed if stable for at least 1 week prior to study Greater than 3rd percentile weight for height

PRIOR CONCURRENT THERAPY: Biologic therapy: More than 6 months since prior bone marrow transplantation More than 1 week since prior growth factor(s) Chemotherapy: At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas) and recovered Endocrine therapy: Concurrent dexamethasone allowed if dose stable for at least 1 week prior to study Radiotherapy: More than 3 months since prior craniospinal irradiation greater than 24 Gy More than 3 months since prior total body irradiation More than 2 weeks since prior focal irradiation to symptomatic metastatic sites No prior stereotactic radiosurgery Concurrent total body irradiation allowed Surgery: See Radiotherapy Other: No other concurrent anticancer or experimental drug therapy Concurrent anticonvulsant drugs allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2000-08; Primary Completion 2003-07 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Toxicities of SU5416 in children and adolescents with refractory CNS malignancies
Dose limiting toxicities of SU5416 in children and adolescents receiving enzyme inducing anticonvulsant drugs and in those not receiving enzyme inducing anticonvulsant drugs | Six weeks
Pharmacokinetics of SU5416 and the effects of enzyme inducing anticonvulsant drugs on the pharmacokinetics

SECONDARY OUTCOMES:
Tumor response to SU5416

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Kieran, MD, PhD, Study Chair — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Kieran MW, Supko JG, Wallace D, Fruscio R, Poussaint TY, Phillips P, Pollack I, Packer R, Boyett JM, Blaney S, Banerjee A, Geyer R, Friedman H, Goldman S, Kun LE, Macdonald T; Pediatric Brain Tumor Consortium. Phase I study of SU5416, a small molecule inhibitor of the vascular endothelial growth factor receptor (VEGFR) in refractory pediatric central nervous system tumors. Pediatr Blood Cancer. 2009 Feb;52(2):169-76. doi: 10.1002/pbc.21873. PMID 19065567